CLINICAL TRIAL: NCT06903169
Title: Understanding End User Preferences for Hand Hygiene Enabling Technologies in Urban and Peri-Urban Lusaka Zambia
Acronym: HHET
Status: Completed | Type: Observational
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: HHET
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Handwashing
Keywords: handwashing facility attributes; handwashing facility ranking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Adult Men: Focus group of adult men
- Adult Women: Focus Group of Adult Women
- Elderly > 65 Years: Focus groups of Elderly above 65 years of age
- Caregivers of Under5: Focus groups of Caregivers of children under five (5)

SUMMARY:
The goal of this study is to explore the perceived attributes, acceptability, and use of various improved handwashing facility designs.

The study aimed to establish what are the characteristics of handwashing facilities (attributes) that are prioritized among various groups of potential end users and how do existing improved HWF designs rank according to these preferences? Also how acceptable are promising HWF designs among multiple groups of potential end users in a real-world setting, how do potential users adapt and modify existing HWF for use in their homes.

ELIGIBILITY:
Inclusion Criteria:

* Living within the designated study area
* Meeting category requirements (i.e adult male, adult women, caregivers of under 5 or elderly (>65)

Exclusion Criteria:

* Not from within designated area
* Less than 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will be based in two peri urban communities located in the western part of Lusaka, George and Matero compounds. George and Matero compounds located geographically next to each other have over 320,000 residents with the majority of residents accessing water from water kiosks that are managed by the local council. Some residents still access water from shallow wells that are generally heavily contaminated and polluted.
  Matero and George compounds are characterized by dense, informal settlement patterns, where housing is unplanned and access to WASH is an ongoing challenge. Water supply from the municipality is largely provided through communal boreholes accessed during limited times in a day at a minimal fee. Where affordability is a challenge, residents often resort to using unprotected shallow wells as their main source of water. During the rainy season flooding is common because of unplanned housing and poor drainage systems. Residents mostly rely o
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Attribute Identification | Same day
  Determine the attributes of handwashing facilities that are important to end users using focus group discussions
Handwashing facility ranking | Same day
  Ranking of handwashing facilities based on attributes identified by end users

CONTACTS AND LOCATIONS:
Locations (1):
- George Health Centre, Lusaka, Lusaka Province, Zambia